CLINICAL TRIAL: NCT05838872
Title: Comparative, Controlled Study to Evaluate the Clinical Accuracy and Usability Performance of the Minuteful - Kidney Urine Analysis Test System Conducted by Lay Users
Brief Title: Evaluation of the Accuracy and Usability of the Minuteful - Kidney Urine Analysis Test System in the Lay User Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACR-US-MCU-SUP
Record Dates: First submitted 2023-04-15; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Albuminuria; Chronic Kidney Diseases; Diabetes; Hypertension
MeSH Terms: conditions — Albuminuria; Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Minuteful - Kidney Urine Analysis Test System (Experimental)
  Interventions: Device: Minuteful - Kidney Urine Analysis Test System

INTERVENTIONS:
Device: Minuteful - Kidney Urine Analysis Test System — Urine samples were collected and tested by a lay user, using the Minuteful - Kidney test device. The lay user test results were compared to the results obtained by testing the same urine sample on the comparison device, the URiSCAN Optima.
  Other Names: Minuteful - Kidney; Minuteful - Kidney Test Device; ACR | U.S. Urine Analysis Test System

SUMMARY:
The purpose of this study was to collect additional performance and clinical data on the Minuteful - Kidney test device (previously "ACR | U.S. Urine Analysis Test System"), following the original data collection (NCT04626271).

This method comparison and usability study was designed to evaluate the agreement levels of the Minuteful - Kidney Test with the comparator device (URiSCAN Optima) as well as the device's usability including the lay user's ability to understand and implement the device instructions. It also evaluates the ease of use of the device under actual use conditions in a simulated home environment.

DETAILED DESCRIPTION:
Eligible subjects meeting the inclusion criteria were recruited at the designated site by the study personnel. Following subject consent, the Minuteful - Kidney test kit, in its original packaging, along with the Minuteful - Kidney smartphone application were provided to the subject in a simulated home- use environment. All subjects were requested to follow the in-app instructions to complete the test, without any guidance from the study staff before, during or after testing. After each subject completed the test, the urine sample was tested by a professional user at the clinical site on the URiSCAN Optima device. Each urine sample was tested twice: once using the Minuteful - kidney test by the lay user and once using the comparator device (URiSCAN Optina) by the professional user.

To evaluate the usability of the device, study staff on-site were asked to observe and document the user performance on key tasks in the study flow as well as information regarding the user behavior while performing the test. Subjects were also asked to answer a usability post-test questionnaire.

ELIGIBILITY:
Inclusion Criteria:

A) Males and Females 18-80 years of age

B) Subjects with a known, well-established medical condition and/or risk factor for kidney damage, that can potentially present as an abnormal concentration of urine albumin:

* Diabetes (Type I/Type II, or Gestational Diabetes)
* High Blood Pressure (i.e., Hypertension)
* Cardiovascular Diseases
* Family History of Kidney Disease
* History of Acute Kidney Injury (AKI)

C) Or; subjects with other medical conditions and/or risk factors that impact kidney function:

* Dyslipidemia
* Heavy smoking
* Obesity
* Inherited kidney disease (e.g. Polycystic kidney disease)
* Prolonged obstruction of the urinary tract from different conditions (e.g. enlarged prostate)
* Malignancies
* Recurrent kidney infections
* Other relevant conditions

D) Subjects who are able to use both hands

E) Subjects who are familiar with the use of a smartphone

F) Subjects who are capable of comprehending and following instructions in English

Exclusion Criteria:

A) Subjects with a major cognitive impairment (e.g.: dementia, memory loss, severe mental disorder)

B) Subjects who are not able to collect urine in a receptacle

C) Subjects who are visually impaired (i.e., cannot read the user manual)

D) Any additional reason that disqualifies the subject from participating in the study according to the study physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Accuracy Evaluation: The Degree of Agreement (%) of the Minuteful - Kidney Urine Analysis Test System as Compared to the Comparator Device | 10 months
  The primary objective of the study is to evaluate the % exact match (percent agreement) and the % ±1 block match (percent agreement) of Minuteful - kidney test (tested by the lay user) compared to the URiSCAN Optima Urine Analyzer (the comparator device, tested by a healthcare professional user), for all reported values (blocks).

SECONDARY OUTCOMES:
Usability Evaluation: User Performance Analysis | 10 months
  The usability of the Minuteful - Kidney Urine Analysis Test System will be determined by evaluating the percentage of study subjects able to perform all required steps and successfully complete the test given only the instructions and training materials provided. In addition, each subject was asked to complete a post test questionnaire to assess the device ease of use by rating the various test steps on a scale of 1 to 5, with 5 being the easiest ("very easy") and 1 the hardest ("very hard"). This questionnaire also included understanding questions in a multiple-choice, quiz-like format, to assess the participants' understanding of essential information and key test procedures in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- AccuMed research associates, Garden City, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT05838872/Prot_SAP_000.pdf